CLINICAL TRIAL: NCT02275663
Title: Phase 2 Study of 5 Days Azacytidine Priming Prior to Fludarabine, Cytarabine and Granulocyte-Colony Stimulating Factor (G-CSF) Combination for Patients With Relapsed or Refractory AML
Brief Title: Azacytidine Plus FLAG for Relapsed or Refractory AML
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Ibraheem Motabi, Consultant, Hematology and BMT, King Fahad Medical City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KFMC-AML01
Record Dates: First submitted 2014-10-20; First posted 2014-10-27 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: relapsed AML; refractory AML; azacytidine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; fludarabine; Cytarabine; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azacytidine plus FLAG (Experimental): Azacytidine 75 mg/m2 = mg IV in 100 ml Normal Saline (NS) over 30 minutes on days -5 t0 -1
  G-CSF 5 mcg/kg subcut on days 0 to + 6
  Fludarabine 30mg/m² in 100ml NS IV daily over 30min., on Days +1 to +5
  Cytarabine 2gm/m² = 500ml NS IV daily over 4h, on Days +1 to +5 Start 4h after completion of fludarabine infusion.
  Interventions: Drug: Azacytidine; Drug: Fludarabine; Drug: Cytarabine; Drug: Filgrastim

INTERVENTIONS:
Drug: Azacytidine
  Other Names: vidaza
Drug: Fludarabine
Drug: Cytarabine
Drug: Filgrastim — G-CSF

SUMMARY:
The purpose of this phase 2 study is to test the efficacy of azacytidine given prior to fludarabine, cytarabine, and G-CSF for the treatment of relapsed or refractory acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16 to 60
2. Patients with a diagnosis of relapse or refractory AML (≥ 20% blast in bone marrow).
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤2
4. Patients must have preserved organ function as defined below:

   * Creatinine ≤ 1.5 mg/dl
   * Total bilirubin ≤ 1.5x upper limit of the normal
   * Alanine aminotransferase (ALT) ≤ 2x upper limit of the normal
   * Left ventricular ejection fraction (LVEF) ≥ 45%

Exclusion Criteria:

1. Patients with a diagnosis of acute promyelocytic leukemia (AML -M3)
2. Pregnant women
3. Patients previously treated with fludarabine are allowed to participate.
4. Patients with Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
complete response rate | 6 weeks
  bone marrow blast <5% with complete neutrophil (>1000/ul) and platelets (>100,000/ul) recovery

SECONDARY OUTCOMES:
leukemia free survival | 1-3 years
  from time of complete remission to time of relapse or death
overall survival | 1-3 yeears
  from date of enrolment to date of death
one year leukemia free survival | 1 year
  probability of leukemia free survival at one year of enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Ibraheem H Motabi, MD, Principal Investigator — King Fahad Medical City
Locations (1):
- King Fahad Medical City, Riyadh, Riyadh Region, Saudi Arabia